CLINICAL TRIAL: NCT03787446
Title: Positron Emission Tomography (PET) Imaging Study in Relapsing-Remitting and Primary-Progressive Multiple Sclerosis (MS): Correlations With Advanced MRI in MS
Brief Title: PET Study in Multiple Sclerosis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of British Columbia (Other)
Collaborators: Hoffmann-La Roche (Industry)
Responsible Party: Principal Investigator, Robert Carruthers, Principal Investigator, University of British Columbia
Other Study IDs: H18-02393
Record Dates: First submitted 2018-12-19; First posted 2018-12-26 (Actual); Last update posted 2019-04-22 (Actual); Status verified 2019-04

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Multiple Sclerosis (MS) patients: 3 Primary Progressive MS patients on no disease modifying therapy and 3 Relapsing-Remitting MS patients on no disease modifying therapy
- Healthy Controls (HC): 3 Healthy volunteers aged between 18-60 years of age

SUMMARY:
While both conventional and advanced MRI techniques offer important insights into MS pathophysiology, important aspects of this inflammatory disorder are undetectable with existing MRI technology. In Multiple Sclerosis (MS), there is growing interest in PET as an imaging modality that can increase the investigator's understanding of the disease processes and may add to an understanding of MS phenotype, particularly when combined with advanced MRI techniques such as myelin water imaging.

DETAILED DESCRIPTION:
This is an exploratory study. PBR28 PET scan is new, promising and exploratory endpoints in MS clinical trials, making sample size estimation difficult.

A separate pre-screening consent form will be issued for the TSPO rs6971 polymorphism and eGFR blood samples, a separate pre-screening step. Eligible participants, according to their TSPO rs6971 polymorphism will be presented a separate study consent form to continue into the clinical trial.

Study Assessments include 1 PET scan, 1 MRI scan, OCT, EDSS exam, physical exam, cognitive questionnaires, etc.

ELIGIBILITY:
Inclusion Criteria:

* Subjects diagnosed with Multiple Sclerosis according to the 2010 McDonald criteria or otherwise in the opinion of the investigator (including relapsing-remitting and primary-progressive).
* Aged 18 to 60 years.
* Mixed affinity binder according to rs6971 TSPO polymorphism1.
* Creatinine clearance over 60 mL/min*). * Blood result valid up to 3 months prior to the MRI scan.

Exclusion Criteria:

* Low and high affinity binders according to rs6971 TSPO polymorphism
* Subject pregnant or breastfeeding.
* Subjects with a Body Mass Index (BMI) >35kg/m³.
* Hospitalization within 1 month of screening visit.
* Medical history or current heart failure
* Medical history or current pulmonary failure
* Current or Historical Drug or alcohol abuse in the opinion of the investigator.
* Regular use of anti-inflammatory agents (more than once a week use of aspirin, NSAIDS, Steroids, immunomodulating drugs), unless patient is able to washout from anti-inflammatory drugs 2 weeks prior to PBR PET scan.
* Neurological disorder other than MS, including Brain Trauma, stroke, Parkinson disease, Alzheimer disease, encephalitis.
* Subjects with a history of radiation treatment or other high amounts of radiation exposure in the opinion of the investigator.
* Subjects with a history of metastatic cancer including solid tumors and hematological malignancies, except basal cell, in situ squamous cell carcinoma of the skin, and in situ carcinoma of the cervix or the uterus that have been excised with clear margins.
* Inability to tolerate lying supine for the duration of the MRI and PET scan.
* Claustrophobia.
* Current use of MS drugs as described by the list of prohibited medications.

Exclusion specific to MRI (All MRI specific criteria is subject to conditions posed by the MRI technologist or radiologist):

* Known or suspected piece of metal in eye(s)
* Irremovable piercing or recent tattoos in the last 6 weeks
* Cardiac pacemakers, wires or defibrillator
* Artificial heart valve
* Brain aneurysm clip
* Electrical stimulator for nerves or bones
* Deep brain stimulator
* Implanted drug infusion pump
* Coil, catheter, or filter in any blood vessel
* Orthopedic hardware (artificial joint, plate, screws) inserted within the last 6 weeks
* Surgery within the last 6 weeks
* Harrington rod for scoliosis
* Other metallic prosthesis
* Any metal fragments, Shrapnel, bullets, or metal prosthesis
* Irremovable dentures, braces or retainer(s)
* IUDs containing metal
* Previous surgery of the brain, eyes, ears, breast, chest, heart, or spine in the opinion of the investigator and MRI technician(s)

Exclusion specific to OCT:

* Medical history of Macular degeneration
* Degenerative and/or symptomatic Retinopathy
* Medical history of Glaucoma
* Medical history of Amblyopia with vision loss
* Medical history of Diabetes

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: 3 untreated RRMS, 3 untreated PPMS and 3 healthy controls
Sampling Method: Probability Sample
Enrollment: 9 (Estimated)
Dates: Start 2019-03-26 (Actual); Primary Completion 2020-03 (Estimated); Study Completion 2020-09 (Estimated)

PRIMARY OUTCOMES:
Whole Brain PBR28 binding | January 2020
  To show an increase in 11C-PBR28 binding in all sub-types of MS compared to healthy controls.

SECONDARY OUTCOMES:
Myelin Water Imaging by MRI | January 2020
  To quantitatively measure the brain levels of water located within myelin
Optical Coherence Tomography | January 2020
  To correlate brain levels of inflammation measured by 11C-PBR28 with Retinal Nerve Fiber Layer (RNFL) thickness on Optical Coherence Tomography (OCT).
MS Spectroscopy | January 2020
  To correlate brain levels of inflammation and myelin measured by PET with cognitive dysfunction in MS patients.

CONTACTS AND LOCATIONS:
Overall Officials: Robert L Carruthers, MD, Principal Investigator — MS Clinical Trials Group
Locations (1):
- UBC MS & NMO Clinical Trials Group, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No